CLINICAL TRIAL: NCT07263477
Title: A Study on the Relationship of Interleukin-7 Receptor Gene Polymorphisms With the Risk of Crohn's Disease Onset and the Efficacy of Infliximab
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-01-228
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Crohn Disease (CD)
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Extract whole genome DNA from peripheral blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CD patients: Some CD patients received intravenous injection of IFX (5mg/kg) at weeks 0, 2, and 6, followed by intravenous injection of the same dose of IFX every 8 weeks to maintain treatment.
  Interventions: Biological: Infliximab
- normal control: no biological agents treatment

INTERVENTIONS:
Biological: Infliximab — Intravenous injection of IFX (5mg/kg) at weeks 0, 2, and 6, followed by intravenous injection of the same dose of IFX every 8 weeks to maintain treatment.
  Groups: CD patients

SUMMARY:
From January 2020 to May 2025, 303 CD patients and 514 normal controls were retrospectively collected from Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. Our study aimed to explore the the relationship of interleukin-7 receptor (IL-7R) gene polymorphisms with the risk of Crohn's disease (CD) onset, the clinicopathological features of CD and the efficacy of infliximab (IFX) therapy.

DETAILED DESCRIPTION:
From January 2020 to May 2025, 303 CD patients and 514 normal controls were retrospectively collected from Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University. Our study aimed to explore the the relationship of interleukin-7 receptor (IL-7R) gene polymorphisms with the risk of Crohn's disease (CD) onset, the clinicopathological features of CD and the efficacy of infliximab (IFX) therapy. Multiple polymerase chain reaction ligase detection technology was used to detect the genotype of IL-7R (rs6897932, rs1494555, rs1494558). According to the Montreal CD classification criteria, patients were divided into different subgroups. The Crohn's Disease Activity Index (CDAI) is used to evaluate clinical activity, while the Simplified Crohn's Disease Endoscopic Score (SES-CD) is used to assess endoscopic activity.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed CD based on comprehensive clinical, colonoscopy, histopathological, laboratory, and radiographic examination results

Exclusion Criteria:

* rheumatoid arthritis, systemic lupus erythematosus, intestinal tuberculosis, ischemic enteritis, radiation enteritis, tumors, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There was no statistically significant difference in the gender ratio, average age, and proportion of smokers between CD group and normal control group. All study subjects are from the Zhejiang Han population who are not related by blood
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Genotypes of IL-7R | Baseline
  multiplex polymerase chain reaction-ligase detection reaction technique

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No